CLINICAL TRIAL: NCT04131959
Title: Ticagrelor CytoSorb Hemoadsorption (TISORB): Prospective, Open, Multi-center, Single-arm Study to Demonstrate the Feasibility of the CytoSorb® 300 mL Device to Remove Ticagrelor During Cardiopulmonary Bypass in Patients on Ticagrelor Undergoing Emergent or Urgent Cardiothoracic Surgery
Brief Title: Ticagrelor CytoSorb Hemoadsorption
Acronym: TISORB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stalled study execution from the impact of the COVID-19 pandemic on the UK NHS
Sponsor: CytoSorbents, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-002; IRAS project ID 264064 (Other: UK Integrated Research Approval System (IRAS))
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Emergent Cardiothoracic Surgery; Bleeding; Drug Removal
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: Prospective, open, multi-center, single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Pharmacodynamic population (Experimental): Single arm
  Interventions: Device: CytoSorb 300 mL device

INTERVENTIONS:
Device: CytoSorb 300 mL device — Intra-operative CytoSorb hemoadsorption of ticagrelor during cardiopulmonary bypass

SUMMARY:
TISORB is a study to show that the CytoSorb device removes ticagrelor from blood during surgery in patients who need emergency surgery on their heart. The hypothesis of TISORB is that removal of ticagrelor by the CytoSorb device during surgery will decrease the risk for surgical bleeding from ticagrelor.

ELIGIBILITY:
Inclusion Criteria:

Cardiothoracic surgery requiring cardiopulmonary bypass ≤ 48 hours following the last dose of ticagrelor.

Exclusion Criteria:

Any cardiothoracic surgery > 48 hours after last dose of ticagrelor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Clutton-Brock, MB, ChB, Principal Investigator — NIHR Trauma Management, MedTech Cooperative
Locations (8):
- United Kingdom (8):
  - Queen Elizabeth Hospital, Birmingham, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Harefield Hospital, Harefield, England
  - Manchester Royal Infirmary, Manchester, England
  - Northern General Hospital, Sheffield, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Royal Infirmary of Edinburgh, Edinburgh, Scotland
  - Golden Jubilee National Hospital, Glasgow, Scotland

RESULTS

PARTICIPANT FLOW:
Groups:
- CytoSorb 300 mL Device Treatment Population: Single arm
Period: Overall Study
Arm/Group | CytoSorb 300 mL Device Treatment Population
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CytoSorb 300 mL Device Treatment Population
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 5
Study patient with last dose of Ticagrelor within 48 hours of surgery [Count of Participants; unit: Participants] | 5

OUTCOME MEASURES:

1. Primary Outcome: Primary Pharmacodynamic Endpoint
Description: Change in platelet reactivity as measured by ADPtest on the Multiplate Analyzer immediately before and after cardiopulmonary bypass. The unit of measure is Aggregation Units (AU).
Time Frame: Immediately before and after cardiopulmonary bypass
Measure: Mean (Standard Deviation); unit: Aggregation Units (AU)
Arm/Group | CytoSorb 300 mL Device Treatment Population
Number analyzed (Participants) | 5
Aggregation Units (AU) | 7 (8)

2. Primary Outcome: Primary Pharmacokinetic Endpoint
Description: Percent change in ticagrelor blood concentration immediately before and after cardiopulmonary bypass.
Time Frame: Immediately before and after cardiopulmonary bypass
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Pharmacodynamic Population
Number analyzed (Participants) | 5
Percent change | 63 (12)

ADVERSE EVENTS:
Time Frame: Up to 30 days after surgery
Arm/Group | CytoSorb 300 mL Device Treatment Population
All-Cause Mortality (participants affected / at risk) | 2/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CytoSorb 300 mL Device Treatment Population (N=5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT04131959/Prot_SAP_001.pdf